CLINICAL TRIAL: NCT05310604
Title: Early Detection of Primary Antibody Deficiencies in Primary Care Facilities by an Algorithm Driven Selection of Serologic Testing in Individuals at Risk.
Acronym: GP-PAD II
Status: Completed | Type: Observational
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, Helen L Leavis, Principal Investigator, Clinical Immunologist (MD, PhD), UMC Utrecht
Other Study IDs: NL74944.041.20
Record Dates: First submitted 2022-03-25; First posted 2022-04-05 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Primary Antibody Deficiencies
MeSH Terms: conditions — Primary Immunodeficiency Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Blood withdrawal — Single blood withdrawal for determination of immunoglobulin levels

SUMMARY:
Rationale: Primary antibody deficiencies (PAD) encompass a group of rare heterogeneous diseases. The clinical presentation may vary widely, including infectious and autoimmune symptoms and increased risk of malignancy. Due to the rarity of the diseases and this wide array of symptoms there is often a delay in diagnosis, of up to 12 years on average1-4. Timely diagnosis of PAD reduces morbidity, mortality and health care costs as effective therapies are available. The currently available screening systems for the broader group of primary immunodeficiencies (PID) have been shown to have poor diagnostic performance5-10 and are time consuming. We have thus developed an algorithm to screen patient records in a primary care setting for risk factors specifically for PAD. Patients with a high risk may undergo a laboratory assessment and referral if necessary, thus reducing the diagnostic delay of PAD. The aim of the current study is to validate this algorithm.

Objective:

Main objective: to validate a screening algorithm for PAD in a primary care setting in the Netherlands.

Study design: Mono-centre cohort study based on regular care data

Study population: Primary care patients aged 12-70 years with the 100 highest scores based on our algorithm.

ELIGIBILITY:
Inclusion Criteria:

* Age between 12 and 70 years
* A total algorithm score that is within the highest 0.66% of the algorithm scores within a single general practitioner's clinic
* Signed informed consent
* Did not meet exclusion criteria during manual evaluation of the health care record

Exclusion Criteria:

* Secondary causes of immunodeficiency as registered by ICPC codes for: multiple myeloma, HIV-infection, anorexia nervosa, bulimia, cystic fibrosis.
* The presence of one of the following during manual screening of the health care record: nephrotic syndrome, current systemic chemotherapy and stage 3-4 liver cirrhosis will be excluded. This could not be done by the algorithm as there is no ICPC code available.

Ages: 12 Years to 70 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Primary care patients aged 12-70 years with the 100 highest scores based on our algorithm.
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2022-05-24 (Actual); Primary Completion 2023-02-20 (Actual); Study Completion 2023-02-20 (Actual)

PRIMARY OUTCOMES:
The percentage of high-risk patients with an eventual PAD diagnosis | measurement december 2022

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
A request for access to the IPD can be submitted, which will be reviewed by the research team.

REFERENCES:
- [Derived] Messelink MA, Welsing PMJ, Devercelli G, Marsden JWN, Leavis HL. Clinical Validation of a Primary Antibody Deficiency Screening Algorithm for Primary Care. J Clin Immunol. 2023 Nov;43(8):2022-2032. doi: 10.1007/s10875-023-01575-8. Epub 2023 Sep 16. PMID 37715890
- [Derived] Messelink MA, Berbers RM, van Montfrans JM, Ellerbroek PM, Gladiator A, Welsing PMJ, Leavis H. Development of a primary care screening algorithm for the early detection of patients at risk of primary antibody deficiency. Allergy Asthma Clin Immunol. 2023 May 27;19(1):44. doi: 10.1186/s13223-023-00790-7. PMID 37245042